CLINICAL TRIAL: NCT04659941
Title: Use of BCG Vaccine as a Preventive Measure for COVID-19 in Health Care Workers
Acronym: ProBCG
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Universidade Federal do Rio de Janeiro (Other)
Collaborators: Ministry of Science and Technology, Brazil (Other)
Responsible Party: Principal Investigator, JOSE ROBERTO LAPA E SILVA, MD, MSc, PhD, Universidade Federal do Rio de Janeiro
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 31942220.8.1001.5257
Record Dates: First submitted 2020-12-08; First posted 2020-12-09 (Actual); Last update posted 2023-05-11 (Actual); Status verified 2023-05

CONDITIONS: COVID 19 Vaccine
Keywords: COVID 19; BCG vaccine
MeSH Terms: conditions — COVID-19 | interventions — BCG Vaccine; Sodium Chloride; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- BCG vaccine (Experimental): 0.1 ml of the reconstituted vaccine to be administered intradermally in the lower insertion of the deltoid muscle, preferably on the right side, in only one occasion
  Interventions: Biological: BCG vaccine
- 0.9% sodium chloride (NaCl) saline solution (Placebo Comparator): 0.1 ml of 0.9% NaCl saline solution to be administered intradermally in the lower insertion of the deltoid muscle, preferably on the right side, in only one occasion
  Interventions: Biological: 0.9% sodium chloride (NaCl) saline solution

INTERVENTIONS:
Biological: BCG vaccine — Using aseptic methods, 1 mL of Sterile Water for Injection, is added to one vial of vaccine. Gently swirl the vial until a homogenous suspension is obtained. Avoid forceful agitation which may cause clumping of the mycobacteria. Drop the immunizing dose of 0.1 mL of BCG VACCINE from the syringe and needle onto the cleansed surface of the skin.
  Arms: BCG vaccine
Biological: 0.9% sodium chloride (NaCl) saline solution — A 0.1 ml of 0.9% NaCl saline solution applied intradermally in the lower insertion of the deltoid muscle of the right arm will be used as placebo, except contraindications or impossibilities.
  Arms: 0.9% sodium chloride (NaCl) saline solution

SUMMARY:
The disease promoted by coronavirus (COVID-19) is caused by Severe Acute Respiratory Syndrome (SARS) caused by Coronavirus type 2 (CoV2), being the first cases identified in December 2019 in China after exposure to the animal market in Wuhan city, China. From the first case to the present day, the COVID-19 epidemic has been identified in 185 countries, with the notification of 2,666,154 cases and 186,144 deaths. In Brazil, more than 45,757 cases and 2,906 confirmed deaths by COVID-19 have been confirmed (Visualized on Apr 23 2020). In our country, to date, testing for COVID-19 occurs only in severe cases and few centers offer the service to health care workers, a population at high risk of infection. BCG is a vaccine produced from a live attenuated strain derived from a Mycobacterium bovis isolate and is widely used worldwide as a tuberculosis (TB) vaccine, but there are studies demonstrating non-specific immunotherapeutic mechanisms of this vaccine that signal a possible relationship with the lowest morbidity and mortality associated with COVID-19 infections worldwide. The present study aims to analyze the role of BCG in the prevention of SARS-CoV-2 infection and also in the occurrence of severe forms of COVID-19 in addition to evaluating the immune response mediated by this vaccine in voluntary health care workers.

DETAILED DESCRIPTION:
Study detailed description can be seen on the protocol attached.

ELIGIBILITY:
Inclusion Criteria:

1. Individuals aged 18 ≥, male or female, not infected with SARS-CoV-2
2. Agreement to participate in the study by signing the Free Informed Consent (FIC)
3. Not being pregnant (in case of women able to become pregnant)
4. Have not received a specific vaccine against COVID-19 or, if vaccinated against SARS-CoV-2, have received the complete immunization schedule only with vaccines approved by ANVISA and implemented by the National Immunization Program, (including the second dose) within a minimum of 15 days prior to the date of inclusion in the study
5. If the participant have not received a specific vaccine against COVID-19 approved by ANVISA, be aware and agree to be able to receive them only 15 days after the intervention proposed in this study

Exclusion Criteria:

1. Professionals with a history of SARS-CoV-2 confirmed infection through RT-PCR or who have already presented clinical and molecular diagnosis of COVID-19 prior to the study
2. Individuals who have not underwent confirmatory tests for COVID-19
3. Breastfeeding
4. Individuals with primary or acquired immunodeficiency
5. Individuals affected by malignant neoplasms
6. Patients treated with high-dose corticosteroids (equivalent to the prednisone dose of 20 mg/day or more) for more than two weeks
7. Patients using other immunosuppressive therapies (antineoplastic chemotherapy, radiotherapy, among others)
8. Individuals with autoimmune diseases
9. Dermatological conditions at the vaccine site or generalized
10. Individuals under treatment for active tuberculosis
11. Individuals with a history of previous tuberculosis treatment
12. Individuals with febrile symptoms [body temperature ≥ 37.5 celsius degree (ºC) in the last 48h]
13. Participation in other prevention clinical trials for COVID-19 (vaccines already approved by ANVISA for use by the National Immunization Program are not included in this item)
14. Report of vaccination with live microorganism administered in the month prior to randomization
15. Require that, if another vaccination with live microorganism is required, it is administered in the month following randomisation (If the other live vaccine can be administered on the same day, this exclusion criterion does not apply)
16. Known anaphylactic reaction to any ingredient in BCG vaccine
17. Adverse reaction prior to BCG vaccine [significant local reaction (abscess) or suppurative lymphadenitis]
18. BCG vaccine administered in the last year

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 752 (Estimated)
Dates: Start 2020-10-01 (Actual); Primary Completion 2022-10-01 (Actual); Study Completion 2024-04-01 (Estimated)

PRIMARY OUTCOMES:
Compare the cumulative incidence of SARS-CoV-2 infection | 6 months
  It is estimated that it will take 376 individuals in each of the comparison groups to ensure a statistical power of 85% for the detection of a risk difference of 5%, considering that the 6 months of follow-up, for a type I error of 5%.
Compare the cumulative incidence of severe forms of COVID-19 | 6 months
  With 376 individuals in each of the comparison groups the study will have a statistical power of approximately 75% for the detection of a risk difference of 2%, considering that the control group will have an accumulated incidence of more severe forms of COVID-19 of 2.5% after 6 months of follow-up, for a type I error of 5%.
Assess the BCG vaccine-mediated immune response in health care workers | 6 months
  SARS-CoV2 infection is estimated to occur in approximately 10% of BCG-vaccinated healthcare professionals (experimental group) and in 30% of non-BCG-vaccinated healthcare professionals (placebo group) In this scenario, with the bearing of 372 health professionals in each arm, SARS-CoV2 infection is expected to be detected in 50 BCG-vaccinated professionals and 150 professionals not vaccinated with BCG. For each subgroup (vaccinated and not vaccinated with BCG) it will be possible to identify the predictive biomarkers of infection by comparing infected professionals with those who were not infected with SARS-CoV2.

CONTACTS AND LOCATIONS:
Overall Officials: Fernanda Carvalho de Q Mello, PHD, Principal Investigator — Universidade Federal do Rio de Janeiro
Locations (1):
- Universidade Federal do Rio de Janeiro, Rio de Janeiro, Rio de Janeiro, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Aaby P, Roth A, Ravn H, Napirna BM, Rodrigues A, Lisse IM, Stensballe L, Diness BR, Lausch KR, Lund N, Biering-Sorensen S, Whittle H, Benn CS. Randomized trial of BCG vaccination at birth to low-birth-weight children: beneficial nonspecific effects in the neonatal period? J Infect Dis. 2011 Jul 15;204(2):245-52. doi: 10.1093/infdis/jir240. PMID 21673035
- [Background] Goodridge HS, Ahmed SS, Curtis N, Kollmann TR, Levy O, Netea MG, Pollard AJ, van Crevel R, Wilson CB. Harnessing the beneficial heterologous effects of vaccination. Nat Rev Immunol. 2016 Jun;16(6):392-400. doi: 10.1038/nri.2016.43. Epub 2016 May 9. PMID 27157064
- [Background] Kleinnijenhuis J, Quintin J, Preijers F, Benn CS, Joosten LA, Jacobs C, van Loenhout J, Xavier RJ, Aaby P, van der Meer JW, van Crevel R, Netea MG. Long-lasting effects of BCG vaccination on both heterologous Th1/Th17 responses and innate trained immunity. J Innate Immun. 2014;6(2):152-8. doi: 10.1159/000355628. Epub 2013 Oct 30. PMID 24192057
- [Background] Netea MG, Joosten LA, Latz E, Mills KH, Natoli G, Stunnenberg HG, O'Neill LA, Xavier RJ. Trained immunity: A program of innate immune memory in health and disease. Science. 2016 Apr 22;352(6284):aaf1098. doi: 10.1126/science.aaf1098. Epub 2016 Apr 21. PMID 27102489
- [Background] Channappanavar R, Zhao J, Perlman S. T cell-mediated immune response to respiratory coronaviruses. Immunol Res. 2014 Aug;59(1-3):118-28. doi: 10.1007/s12026-014-8534-z. PMID 24845462
- [Background] Netea MG, Giamarellos-Bourboulis EJ, Dominguez-Andres J, Curtis N, van Crevel R, van de Veerdonk FL, Bonten M. Trained Immunity: a Tool for Reducing Susceptibility to and the Severity of SARS-CoV-2 Infection. Cell. 2020 May 28;181(5):969-977. doi: 10.1016/j.cell.2020.04.042. Epub 2020 May 4. PMID 32437659
- [Background] Ozdemir C, Kucuksezer UC, Tamay ZU. Is BCG vaccination affecting the spread and severity of COVID-19? Allergy. 2020 Jul;75(7):1824-1827. doi: 10.1111/all.14344. Epub 2020 May 12. No abstract available. PMID 32330314
- [Background] Urashima M, Otani K, Hasegawa Y, Akutsu T. BCG Vaccination and Mortality of COVID-19 across 173 Countries: An Ecological Study. Int J Environ Res Public Health. 2020 Aug 3;17(15):5589. doi: 10.3390/ijerph17155589. PMID 32756371
- [Derived] Santos AP, Werneck GL, Dalvi APR, Dos Santos CC, Tierno PFGMM, Condelo HS, Macedo B, de Medeiros Leung JA, de Souza Nogueira J, Malvao L, Galliez R, Aguiar R, Stefan R, Knackfuss SM, da Silva EC, Castineiras TMPP, de Andrade Medronho R, E Silva JRL, Alves RLR, de Moraes Sobrino Porto LC, Rodrigues LS, Kritski AL, de Queiroz Mello FC. The effect of BCG vaccination on infection and antibody levels against SARS-CoV-2-The results of ProBCG: a multicenter randomized clinical trial in Brazil. Int J Infect Dis. 2023 May;130:8-16. doi: 10.1016/j.ijid.2023.02.014. Epub 2023 Feb 24. PMID 36841502

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-09-30): https://cdn.clinicaltrials.gov/large-docs/41/NCT04659941/Prot_SAP_001.pdf
  • Informed Consent Form (2021-09-30): https://cdn.clinicaltrials.gov/large-docs/41/NCT04659941/ICF_002.pdf